CLINICAL TRIAL: NCT06292481
Title: Combine Effects of Brunnstorm Movement Therapy and LLLT on Upper Limb Functioning and Hand Dexterity in Chronic Stroke Patient
Brief Title: Combine Effects of Brunnstorm Movement Therapy and LLLT in Chronic Stroke Patient
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0240
Record Dates: First submitted 2024-01-28; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Chronic Stroke
Keywords: Brunnstorm movement therapy; Hand dexterity; Low-level laser therapy; Stroke
MeSH Terms: conditions — Stroke | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brunnstorm Movement therapy (Experimental): this group received Brunnstorm Movement therapy for 3 to 5 sessions per week, each lasting approximately 30 to 60 minutes for 6 weeks
  Interventions: Other: Brunnstorm movement therapy
- Combined Brunnstorm Movement therapy and low level laser therapy (Experimental): this group received Combined Brunnstorm Movement therapy and low level laser therapy for 3 to 5 sessions per week, each lasting approximately 30 to 60 minutes for 6 weeks
  Interventions: Other: Combined Brunnstorm Movement therapy and low level laser therapy

INTERVENTIONS:
Other: Brunnstorm movement therapy — this group received Brunnstorm Movement therapy for 3 to 5 sessions per week, each lasting approximately 30 to 60 minutes for 6 weeks
  Arms: Brunnstorm Movement therapy
Other: Combined Brunnstorm Movement therapy and low level laser therapy — this group received Combined Brunnstorm Movement therapy and low level laser therapy for 3 to 5 sessions per week, each lasting approximately 30 to 60 minutes for 6 weeks
  Arms: Combined Brunnstorm Movement therapy and low level laser therapy

SUMMARY:
The primary objective of this study is to determine the combined effects of Brunnstorm movement therapy and low level laser therapy on upper limb function in chronic stroke patient.

ELIGIBILITY:
Inclusion Criteria:

* Age range between 40 & 60 years (16)
* Both males and females.
* Combined Effects of Brunnstorm movement therapy and LLLT on Upper limb function Hand dexterity in stroke
* Patient with maximum Grade 1 and 1+ spasticity according to Modified
* Ashworth scale and minimum muscle strength of 1 in the biceps brachii muscle.
* Onset of injury : (1 to 2 years)

Exclusion Criteria:

* Any comorbidity such as malignancy, inflammatory rheumatologic disease, rheumatoid arthritis, ankylosing spondylitis, psoriatic arthritis, lupus erythematosus, etc.
* Have a pacemaker or a history of serious cardiac events or of cardiorespiratory dysfunction.
* Visual impairment
* Any other musculoskeletal disorders of extremity
* Severe cognitive impairment or aphasia leading to difficulty in communication, Participants unwilling to comply with the protocol.

Ages: 40 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Fugle meyer Assessment test | 6th week
Box and block test | 6th week
Nine peg hole test | 6th week
to check Muscle tone | 6th week
  Modified Ashworth Scale
to measure grip Strength | 6th week
  Hand handled dynamometer

CONTACTS AND LOCATIONS:
Overall Officials: Binash Afzal, PHD*, Principal Investigator — Riphah international university lahore campus
Locations (1):
- Govt. Mian Munshi DHQ Teaching hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] das Neves MF, Aleixo DC, Mendes IS, Lima FPS, Nicolau RA, Arisawa EAL, Lopes-Martins RAB, Lima MO. Long-term analyses of spastic muscle behavior in chronic poststroke patients after near-infrared low-level laser therapy (808 nm): a double-blinded placebo-controlled clinical trial. Lasers Med Sci. 2020 Sep;35(7):1459-1467. doi: 10.1007/s10103-019-02920-3. Epub 2019 Dec 10. PMID 31823135
- [Background] da Silva BP, Souza GADS, Filho AADN, Pinto AP, Guimaraes CL, Pereira APC, Neves MFD, Martins PSLL, Lima FPS, Lopes-Martins RAB, Lima MO. Analysis of the effects of low-level laser therapy on muscle fatigue of the biceps brachii muscle of healthy individuals and spastic individuals: Study protocol for a single-center, randomized, double-blind, and controlled clinical trial. Medicine (Baltimore). 2019 Sep;98(39):e17166. doi: 10.1097/MD.0000000000017166. PMID 31574822
- [Background] Azuma RHE, Merlo JK, Jacinto JL, Borim JM, da Silva RA, Pacagnelli FL, Nunes JP, Ribeiro AS, Aguiar AF. Photobiomodulation Therapy at 808 nm Does Not Improve Biceps Brachii Performance to Exhaustion and Delayed-Onset Muscle Soreness in Young Adult Women: A Randomized, Controlled, Crossover Trial. Front Physiol. 2021 Jun 10;12:664582. doi: 10.3389/fphys.2021.664582. eCollection 2021. PMID 34177615
- [Background] Stamborowski SF, de Oliveira Spinelli BM, Lima FPS, Costa DR, de Silveira Souza GA, Lima MO, Lopes Martins RAB. The influence of photobiomodulation on the temperature of the brachial biceps during muscle fatigue protocol. Lasers Med Sci. 2021 Oct;36(8):1741-1749. doi: 10.1007/s10103-021-03360-8. Epub 2021 Jul 13. PMID 34255219
- [Background] Vassao PG, Baldini GS, Vieira KVSG, Balao AB, Pinfildi CE, Campos RMDS, Tucci HT, Renno ACM. Acute Photobiomodulation Effects Through a Cluster Device on Skeletal Muscle Fatigue of Biceps Brachii in Young and Healthy Males: A Randomized Double-Blind Session. Photobiomodul Photomed Laser Surg. 2020 Dec;38(12):773-779. doi: 10.1089/photob.2019.4786. PMID 33332234
- [Background] Harada T, Miyagi M, Izukura H, Endou G, Ushigome N, Tsuruoka H, Mizutani A, Ohshiro T, Ebihara S. The effect of low level laser therapy for pain in major muscles controlling two joints. Laser Ther. 2019 Jun 30;28(2):111-115. doi: 10.5978/islsm.19-OR-07. PMID 32921909